CLINICAL TRIAL: NCT01812252
Title: Initial Cytoreductive Therapy for Myelodysplastic Syndrome Prior to Allogeneic Hematopoietic Cell Transplantation (the ICT-HCT Study)
Brief Title: Chemotherapy in Treating Patients With Myelodysplastic Syndrome Before Donor Stem Cell Transplant
Acronym: ICT-HCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Principal Investigator, Bart Scott, Professor, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2661.00; NCI-2013-00538 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2661; 2661.00 (Other: Fred Hutch/University of Washington Cancer Consortium); RG9215001 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Results first posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-01

CONDITIONS: Chronic Myelomonocytic Leukemia; de Novo Myelodysplastic Syndrome; Myelodysplastic Syndrome; Secondary Myelodysplastic Syndrome
Keywords: myelodysplastic syndrome; chronic myelomonocytic leukemia; bone marrow transplant; hypomethylating agent; induction chemotherapy
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes | interventions — Azacitidine; Decitabine; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (decitabine or azacitidine) (Other): Patients receive decitabine or azacitidine IV or SC per standard of care. Treatment repeats per standard of care, every 28 days for 4 cycles of decitabine or 6 cycles of azacitidine in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine (AZC); Drug: Decitabine; Other: Quality-of-Life Assessment
- Arm B (induction-like chemotherapy regimen) (Other): Patients receive physician choice of standard of care or other experimental protocol using induction-like chemotherapy regimen. No one specific regimen is required. Several regimens are listed in the protocol for example only.
  Interventions: Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Azacitidine (AZC) — Given IV or SC
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; AZACITIDINE; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
  Arms: Arm A (decitabine or azacitidine)
Drug: Decitabine — Given IV or SC
  Other Names: 5-Aza-2'-deoxycytidine; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
  Arms: Arm A (decitabine or azacitidine)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This randomized clinical trial studies different chemotherapies in treating patients with myelodysplastic syndrome before donor stem cell transplant. Giving chemotherapy before a donor stem cell transplant helps stop the growth of cancer cells in the bone marrow, including normal blood-forming cells (stem cells) and cancer cells, and may prevent the myelodysplastic syndrome from coming back after the transplant. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 2 treatment arms.

Arm A: Patients receive decitabine or azacitidine intravenously (IV) or subcutaneously (SC) for 7 days. Treatment repeats every 28 days for 4 cycles of decitabine or 6 cycles of azacitidine in the absence of disease progression or unacceptable toxicity.

Arm B: Patients receive induction-like chemotherapy per standard of care or per experimental protocol. This study does not require a specific chemotherapy regimen for Arm B.

After completion of study treatment, patients are followed up for 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of de novo or secondary myelodysplastic syndrome (MDS), including chronic myelomonocytic leukemia, as defined by the 2008 World Health Organization classification system
* Patients must have measurable disease requiring cytoreduction, defined as a bone marrow myeloblast count >= 5% and < 20% on morphologic examination or by flow cytometry in cases in which adequate morphologic examination is not possible
* Patients must be considered to have an acceptable risk of early mortality with intensive chemotherapy as determined by the attending physician at the time of the initial visit; since the specific therapy within each arm will be determined after randomization, there is no threshold of organ dysfunction or performance status for inclusion
* Considered a potential transplant candidate; the attending/treating physician will determine transplant candidacy at the time of consent
* Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent

Exclusion Criteria:

* A diagnosis of acute promyelocytic leukemia as defined by the 2008 World Health Organization classification system
* Previous treatment for MDS or acute myeloblastic leukemia (AML) with intensive chemotherapy regimen (induction chemotherapy) or hypomethylating agent
* Have any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver, or other organ system that may place the patient at undue risk to undergo treatment
* Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment)
* Females who are pregnant or breastfeeding
* Fertile men and women unwilling to use contraceptive techniques during and for 12 months following treatment
* Any uncontrolled or significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results
* Clinical evidence suggestive of central nervous system (CNS) involvement with MDS unless a lumbar puncture confirms the absence of leukemic blasts in the cerebrospinal fluid (CSF)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-08-19 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bart L. Scott, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (4):
- United States (4):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington

REFERENCES:
- [Background] Greenberg P, Cox C, LeBeau MM, Fenaux P, Morel P, Sanz G, Sanz M, Vallespi T, Hamblin T, Oscier D, Ohyashiki K, Toyama K, Aul C, Mufti G, Bennett J. International scoring system for evaluating prognosis in myelodysplastic syndromes. Blood. 1997 Mar 15;89(6):2079-88. PMID 9058730
- [Background] Gooley TA, Chien JW, Pergam SA, Hingorani S, Sorror ML, Boeckh M, Martin PJ, Sandmaier BM, Marr KA, Appelbaum FR, Storb R, McDonald GB. Reduced mortality after allogeneic hematopoietic-cell transplantation. N Engl J Med. 2010 Nov 25;363(22):2091-101. doi: 10.1056/NEJMoa1004383. PMID 21105791
- [Background] Deeg HJ, Storer B, Slattery JT, Anasetti C, Doney KC, Hansen JA, Kiem HP, Martin PJ, Petersdorf E, Radich JP, Sanders JE, Shulman HM, Warren EH, Witherspoon RP, Bryant EM, Chauncey TR, Getzendaner L, Storb R, Appelbaum FR. Conditioning with targeted busulfan and cyclophosphamide for hemopoietic stem cell transplantation from related and unrelated donors in patients with myelodysplastic syndrome. Blood. 2002 Aug 15;100(4):1201-7. doi: 10.1182/blood-2002-02-0527. PMID 12149198
- [Background] Lim Z, Brand R, Martino R, van Biezen A, Finke J, Bacigalupo A, Beelen D, Devergie A, Alessandrino E, Willemze R, Ruutu T, Boogaerts M, Falda M, Jouet JP, Niederwieser D, Kroger N, Mufti GJ, De Witte TM. Allogeneic hematopoietic stem-cell transplantation for patients 50 years or older with myelodysplastic syndromes or secondary acute myeloid leukemia. J Clin Oncol. 2010 Jan 20;28(3):405-11. doi: 10.1200/JCO.2009.21.8073. Epub 2009 Dec 14. PMID 20008642
- [Background] Warlick ED, Cioc A, Defor T, Dolan M, Weisdorf D. Allogeneic stem cell transplantation for adults with myelodysplastic syndromes: importance of pretransplant disease burden. Biol Blood Marrow Transplant. 2009 Jan;15(1):30-8. doi: 10.1016/j.bbmt.2008.10.012. PMID 19135940
- [Background] Nakai K, Kanda Y, Fukuhara S, Sakamaki H, Okamoto S, Kodera Y, Tanosaki R, Takahashi S, Matsushima T, Atsuta Y, Hamajima N, Kasai M, Kato S. Value of chemotherapy before allogeneic hematopoietic stem cell transplantation from an HLA-identical sibling donor for myelodysplastic syndrome. Leukemia. 2005 Mar;19(3):396-401. doi: 10.1038/sj.leu.2403640. PMID 15674354
- [Background] Scott BL, Storer B, Loken MR, Storb R, Appelbaum FR, Deeg HJ. Pretransplantation induction chemotherapy and posttransplantation relapse in patients with advanced myelodysplastic syndrome. Biol Blood Marrow Transplant. 2005 Jan;11(1):65-73. doi: 10.1016/j.bbmt.2004.10.001. PMID 15625546
- [Background] Yakoub-Agha I, de La Salmoniere P, Ribaud P, Sutton L, Wattel E, Kuentz M, Jouet JP, Marit G, Milpied N, Deconinck E, Gratecos N, Leporrier M, Chabbert I, Caillot D, Damaj G, Dauriac C, Dreyfus F, Francois S, Molina L, Tanguy ML, Chevret S, Gluckman E. Allogeneic bone marrow transplantation for therapy-related myelodysplastic syndrome and acute myeloid leukemia: a long-term study of 70 patients-report of the French society of bone marrow transplantation. J Clin Oncol. 2000 Mar;18(5):963-71. doi: 10.1200/JCO.2000.18.5.963. PMID 10694545
- [Background] Estey E, de Lima M, Tibes R, Pierce S, Kantarjian H, Champlin R, Giralt S. Prospective feasibility analysis of reduced-intensity conditioning (RIC) regimens for hematopoietic stem cell transplantation (HSCT) in elderly patients with acute myeloid leukemia (AML) and high-risk myelodysplastic syndrome (MDS). Blood. 2007 Feb 15;109(4):1395-400. doi: 10.1182/blood-2006-05-021907. Epub 2006 Oct 12. PMID 17038533
- [Background] De Padua Silva L, de Lima M, Kantarjian H, Faderl S, Kebriaei P, Giralt S, Davisson J, Garcia-Manero G, Champlin R, Issa JP, Ravandi F. Feasibility of allo-SCT after hypomethylating therapy with decitabine for myelodysplastic syndrome. Bone Marrow Transplant. 2009 Jun;43(11):839-43. doi: 10.1038/bmt.2008.400. Epub 2009 Jan 19. PMID 19151791
- [Background] Field T, Perkins J, Huang Y, Kharfan-Dabaja MA, Alsina M, Ayala E, Fernandez HF, Janssen W, Lancet J, Perez L, Sullivan D, List A, Anasetti C. 5-Azacitidine for myelodysplasia before allogeneic hematopoietic cell transplantation. Bone Marrow Transplant. 2010 Feb;45(2):255-60. doi: 10.1038/bmt.2009.134. Epub 2009 Jun 22. PMID 19543327
- [Background] Lubbert M, Bertz H, Ruter B, Marks R, Claus R, Wasch R, Finke J. Non-intensive treatment with low-dose 5-aza-2'-deoxycytidine (DAC) prior to allogeneic blood SCT of older MDS/AML patients. Bone Marrow Transplant. 2009 Nov;44(9):585-8. doi: 10.1038/bmt.2009.64. Epub 2009 Apr 13. PMID 19363531
- [Background] Gerds AT, Gooley TA, Estey EH, Appelbaum FR, Deeg HJ, Scott BL. Pretransplantation therapy with azacitidine vs induction chemotherapy and posttransplantation outcome in patients with MDS. Biol Blood Marrow Transplant. 2012 Aug;18(8):1211-8. doi: 10.1016/j.bbmt.2012.01.009. Epub 2012 Jan 16. PMID 22252125
- [Background] Fenaux P, Mufti GJ, Hellstrom-Lindberg E, Santini V, Finelli C, Giagounidis A, Schoch R, Gattermann N, Sanz G, List A, Gore SD, Seymour JF, Bennett JM, Byrd J, Backstrom J, Zimmerman L, McKenzie D, Beach C, Silverman LR; International Vidaza High-Risk MDS Survival Study Group. Efficacy of azacitidine compared with that of conventional care regimens in the treatment of higher-risk myelodysplastic syndromes: a randomised, open-label, phase III study. Lancet Oncol. 2009 Mar;10(3):223-32. doi: 10.1016/S1470-2045(09)70003-8. Epub 2009 Feb 21. PMID 19230772
- [Background] Lowenberg B, Ossenkoppele GJ, van Putten W, Schouten HC, Graux C, Ferrant A, Sonneveld P, Maertens J, Jongen-Lavrencic M, von Lilienfeld-Toal M, Biemond BJ, Vellenga E, van Marwijk Kooy M, Verdonck LF, Beck J, Dohner H, Gratwohl A, Pabst T, Verhoef G; Dutch-Belgian Cooperative Trial Group for Hemato-Oncology (HOVON); German AML Study Group (AMLSG); Swiss Group for Clinical Cancer Research (SAKK) Collaborative Group. High-dose daunorubicin in older patients with acute myeloid leukemia. N Engl J Med. 2009 Sep 24;361(13):1235-48. doi: 10.1056/NEJMoa0901409. PMID 19776405
- [Background] Pautas C, Merabet F, Thomas X, Raffoux E, Gardin C, Corm S, Bourhis JH, Reman O, Turlure P, Contentin N, de Revel T, Rousselot P, Preudhomme C, Bordessoule D, Fenaux P, Terre C, Michallet M, Dombret H, Chevret S, Castaigne S. Randomized study of intensified anthracycline doses for induction and recombinant interleukin-2 for maintenance in patients with acute myeloid leukemia age 50 to 70 years: results of the ALFA-9801 study. J Clin Oncol. 2010 Feb 10;28(5):808-14. doi: 10.1200/JCO.2009.23.2652. Epub 2010 Jan 4. PMID 20048183

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at 3 academic medical centers between April 2013 to March 2022. The first participant was enrolled on August 19, 2013 and the last participant was enrolled in September 24, 2021.
Pre-assignment Details: This study is a multi-center, open-label randomized study of intensive chemotherapy versus hypomethylating agent-based therapy as the initial pre-transplant cytoreductive therapy in patients with myelodysplastic syndrome.
  Patients will be randomized to receive treatment with either hypomethylating agent therapy or intensive chemotherapy; they will not receive both.
Period: Overall Study
Arm/Group | Arm A (Decitabine or Azacitidine) | Arm B (Induction-like Chemotherapy Regimen)
Started | 25 | 25
Completed | 6 | 10
Not Completed | 19 | 15
Not completed — Persistent Disease | 1 | 0
Not completed — Not transplanted | 11 | 11
Not completed — Transplanted died prior to 18-months post-transplant follow-up | 5 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Screen Failure | 1 | 0

BASELINE CHARACTERISTICS:
Population: Eligible patients will be randomized in a 1:1 fashion. The primary outcome will be analyzed on an intention-to-treat basis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Decitabine or Azacitidine) | Arm B (Induction-like Chemotherapy Regimen) | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 14 | 27
  >=65 years | 12 | 11 | 23
Age, Continuous [Mean (Full Range); unit: years] | 59.9 [27.3 to 78.4] | 60.7 [31.9 to 73.6] | 60.3 [27.3 to 78.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 17 | 15 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 25 | 24 | 49
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 23 | 21 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Failure-free Survival (Failure Defined as Death or Relapse)
Description: 18-month failure-free survival (failure defined as death or relapse).
Time Frame: 18 months
Population: Number of subjects enrolled and randomized in each arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Decitabine or Azacitidine) | Arm B (Induction-like Chemotherapy Regimen)
Number analyzed (Participants) | 25 | 25
Participants | 6 | 10

2. Secondary Outcome: Quality of Life Will be Assessed Using the European Organization for Research and Treatment of Cancer Quality of Life (QoL) Questionnaire (EORTC QLQ-C30) Questionnaire.
Description: The European Organization for Research and Treatment of Cancer Quality of Life (EORTC QLQ-C30) (version 3) is a 30-item cancer-specific questionnaire for measuring the health-related quality of life (QOL) in cancer patients. It includes five functioning scales (physical, PF; role, RF; cognitive, CF; emotional, EF; and social, SF), three symptom scales (fatigue, FA; pain, PA; and nausea and vomiting, NV), a global health status/QOL scale (GL), and six single items (dyspnea, appetite loss, sleep disturbance, constipation, diarrhea, and financial impact of the disease and treatment). All items employ a 4-point Likert scale, ranging from 1 (not at all) to 4 (very much) with lower scores representing a better outcome and higher scores a worse outcome; with the exception of two items in the GL scale, which use 7-point scales (1=very poor to 7=excellent) lower scores representing a worse outcome and higher score representing a better outcome.
Time Frame: EORTC QLQ-C30 questionnaire will be collected at screening, after completion of therapy (HMA 4-6 month, and up to 6 months for induction-like chemotherapy) just prior to stem cell infusion and 100 (± 14) days after stem cell infusion (HSCT).
Population: The QLQ-C30 is a validated and widely used questionnaire to assess QOL in cancer patients. For Arm A (Azacitidine or Decitabine) only 22 subjects submitted EORTC QLQ-C30 at screening; 14 subjects completed EORTC QLQ-C30 at pre-transplant and 10 subjects post-transplant. For Arm B (induction chemo) 25 subjects submitted EORTC QLQ-C30 at screening; 13 subjects completed QLQ-C30 at pre-transplant and 10 subjects post-transplant. Scores for each question and timepoints were averaged to obtain mean.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Arm A (Azacitidine or Decitabine): Patients receive decitabine or azacitidine IV or SC per standard of care. Treatment repeats per standard of care, every 28 days for 4 cycles of decitabine or 6 cycles of azacitidine in the absence of disease progression or unacceptable toxicity.
  Azacitidine (AZC): Given IV or SC
  Decitabine: Given IV or SC
- Arm B (Induction Like Chemotherapy): Patients receive physician choice of standard of care or other experimental protocol using induction-like chemotherapy regimen. No one specific regimen is required. Several regimens are listed in the protocol for example only.
Arm/Group | Arm A (Azacitidine or Decitabine) | Arm B (Induction Like Chemotherapy)
Number analyzed (Participants) | 25 | 25
score on a scale
  EORTCQLQ-C30 at Screening 1. Do you have any trouble doing strenuous activities?: number analyzed (Participants) | 22 | 25
  EORTCQLQ-C30 at Screening 1. Do you have any trouble doing strenuous activities? | 2.27 [1 to 4] | 1.72 [1 to 4]
  EORTCQLQ-C30 at Pre-Transplant 1. Do you have any trouble doing strenuous activities?: number analyzed (Participants) | 14 | 13
  EORTCQLQ-C30 at Pre-Transplant 1. Do you have any trouble doing strenuous activities? | 2.14 [1 to 4] | 2.0 [1 to 4]
  EORTCQLQ-C30 at post-transplant 1. Do you have any trouble doing strenuous activities?: number analyzed (Participants) | 10 | 10
  EORTCQLQ-C30 at post-transplant 1. Do you have any trouble doing strenuous activities? | 2.0 [1 to 4] | 1.81 [1 to 4]
  EORTCQLQ-C30 at Screening 2. Do you have any trouble taking a long walk?: number analyzed (Participants) | 22 | 25
  EORTCQLQ-C30 at Screening 2. Do you have any trouble taking a long walk? | 2.40 [1 to 4] | 1.96 [1 to 4]
  EORTCQLQ-C30 at Pre-transplant 2. Do you have any trouble taking a long walk?: number analyzed (Participants) | 14 | 13
  EORTCQLQ-C30 at Pre-transplant 2. Do you have any trouble taking a long walk? | 1.85 [1 to 4] | 1.83 [1 to 4]
  EORTCQLQ-C30 at Post-transplant 2. Do you have any trouble taking a long walk?: number analyzed (Participants) | 10 | 10
  EORTCQLQ-C30 at Post-transplant 2. Do you have any trouble taking a long walk? | 1.9 [1 to 4] | 1.63 [1 to 4]
  EORTCQLQ-C30 at Screening 3. Do you have any trouble taking a short walk outside of the house?: number analyzed (Participants) | 22 | 25
  EORTCQLQ-C30 at Screening 3. Do you have any trouble taking a short walk outside of the house? | 1.5 [1 to 4] | 1.24 [1 to 4]
  EORTCQLQ-C30 at Pre-transplant 3. Do you have any trouble taking a short walk outside of the house?: number analyzed (Participants) | 14 | 13
  EORTCQLQ-C30 at Pre-transplant 3. Do you have any trouble taking a short walk outside of the house? | 1.42 [1 to 4] | 1.30 [1 to 4]
  EORTCQLQ-C30 at Post-transplant 3.Do you have any trouble taking a short walk outside of the house?: number analyzed (Participants) | 10 | 10
  EORTCQLQ-C30 at Post-transplant 3.Do you have any trouble taking a short walk outside of the house? | 1.1 [1 to 4] | 1.4 [1 to 4]
  EORTCQLQ-C30 at Screening 4. Do you need to stay in bed or a chair during the day?: number analyzed (Participants) | 22 | 25
  EORTCQLQ-C30 at Screening 4. Do you need to stay in bed or a chair during the day? | 1.68 [1 to 4] | 1.66 [1 to 4]
  EORTCQLQ-C30 at Pre transplant 4. Do you need to stay in bed or a chair during the day?: number analyzed (Participants) | 14 | 13
  EORTCQLQ-C30 at Pre transplant 4. Do you need to stay in bed or a chair during the day? | 1.42 [1 to 4] | 1.30 [1 to 4]
  EORTCQLQ-C30 at Post-transplant 4. Do you need to stay in bed or a chair during the day?: number analyzed (Participants) | 10 | 10
  EORTCQLQ-C30 at Post-transplant 4. Do you need to stay in bed or a chair during the day? | 1.45 [1 to 4] | 1.5 [1 to 4]
  EORTCQLQ-C30 at Screening 5. Do you need help with eating, dressing, washing yourself?: number analyzed (Participants) | 22 | 25
  EORTCQLQ-C30 at Screening 5. Do you need help with eating, dressing, washing yourself? | 1.04 [1 to 4] | 1.08 [1 to 4]
  EORTCQLQ-C30 at Pre-transplant 5. Do you need help with eating, dressing, washing yourself?: number analyzed (Participants) | 14 | 13
  EORTCQLQ-C30 at Pre-transplant 5. Do you need help with eating, dressing, washing yourself? | 1 [1 to 4] | 1 [1 to 4]
  EORTCQLQ-C30 at Post-transplant 5. Do you need help with eating, dressing, washing yourself? | 1 [1 to 4] | 1 [1 to 4]
  EORTCQLQ-C30 at Screening 6. Were you limited in doing either your work or other daily activities?: number analyzed (Participants) | 22 | 25
  EORTCQLQ-C30 at Screening 6. Were you limited in doing either your work or other daily activities? | 2.22 [1 to 4] | 1.92 [1 to 4]
  EORTCQLQ-C30 Pre-transplant 6.Were you limited in doing either your work or other daily activities?: number analyzed (Participants) | 14 | 13
  EORTCQLQ-C30 Pre-transplant 6.Were you limited in doing either your work or other daily activities? | 2.07 [1 to 4] | 1.61 [1 to 4]
  EORTCQLQ-C30 Post-Transplant 6.Were you limited in doing either your work/ other daily activities?: number analyzed (Participants) | 10 | 10
  EORTCQLQ-C30 Post-Transplant 6.Were you limited in doing either your work/ other daily activities? | 1.8 [1 to 4] | 1.8 [1 to 4]
  EORTCQLQ-C30 Screening 7.Were you limited in pursing your hobbies or other leisure time activities?: number analyzed (Participants) | 22 | 25
  EORTCQLQ-C30 Screening 7.Were you limited in pursing your hobbies or other leisure time activities? | 2.52 [1 to 4] | 1.88 [1 to 4]
  EORTCQLQ-C30 Pre-transplant 7.Were you limited in pursing your hobbies/other leisure activities?: number analyzed (Participants) | 14 | 13
  EORTCQLQ-C30 Pre-transplant 7.Were you limited in pursing your hobbies/other leisure activities? | 2.07 [1 to 4] | 1.85 [1 to 4]
  EORTCQLQ-C30 Post-transplant 7.Were you limited in pursing your hobbies/other leisure activities?: number analyzed (Participants) | 10 | 10
  EORTCQLQ-C30 Post-transplant 7.Were you limited in pursing your hobbies/other leisure activities? | 1.9 [1 to 4] | 1.8 [1 to 4]
  EORTCQLQ-C30 Screening 8. Were you short of breath?: number analyzed (Participants) | 22 | 25
  EORTCQLQ-C30 Screening 8. Were you short of breath? | 2.22 [1 to 4] | 2 [1 to 4]
  EORTCQLQ-C30 Pre-transplant 8. Were you short of breath?: number analyzed (Participants) | 14 | 13
  EORTCQLQ-C30 Pre-transplant 8. Were you short of breath? | 1.85 [1 to 4] | 1.31 [1 to 4]
  EORTCQLQ-C30 Post-transplant 8. Were you short of breath?: number analyzed (Participants) | 10 | 10
  EORTCQLQ-C30 Post-transplant 8. Were you short of breath? | 1.5 [1 to 4] | 1.33 [1 to 4]
  EORTCQLQ-C30 Screening 9. Have you had pain?: number analyzed (Participants) | 22 | 25
  EORTCQLQ-C30 Screening 9. Have you had pain? | 1.54 [1 to 4] | 1.48 [1 to 4]
  EORTCQLQ-C30 Pre-transplant 9. Have you had pain?: number analyzed (Participants) | 14 | 13
  EORTCQLQ-C30 Pre-transplant 9. Have you had pain? | 1.78 [1 to 4] | 1.46 [1 to 4]
  EORTCQLQ-C30 Post-transplant 9. Have you had pain?: number analyzed (Participants) | 10 | 10
  EORTCQLQ-C30 Post-transplant 9. Have you had pain? | 1.6 [1 to 4] | 1.4 [1 to 4]
  EORTCQLQ-C30 Screening 10. Did you need to rest?: number analyzed (Participants) | 22 | 25
  EORTCQLQ-C30 Screening 10. Did you need to rest? | 2.38 [1 to 4] | 2.16 [1 to 4]
  EORTCQLQ-C30 Pre-transplant 10. Did you need to rest?: number analyzed (Participants) | 14 | 13
  EORTCQLQ-C30 Pre-transplant 10. Did you need to rest? | 2.21 [1 to 4] | 2.15 [1 to 4]
  EORTCQLQ-C30 Post-transplant 10. Did you need to rest?: number analyzed (Participants) | 10 | 10
  EORTCQLQ-C30 Post-transplant 10. Did you need to rest? | 1.9 [1 to 4] | 2.0 [1 to 4]
  EORTCQLQ-C30 Screening 11. Have you had trouble sleeping?: number analyzed (Participants) | 22 | 25
  EORTCQLQ-C30 Screening 11. Have you had trouble sleeping? | 2.0 [1 to 4] | 1.8 [1 to 4]
  EORTCQLQ-C30 Pre-transplant 11. Have you had trouble sleeping?: number analyzed (Participants) | 14 | 13
  EORTCQLQ-C30 Pre-transplant 11. Have you had trouble sleeping? | 2.35 [1 to 4] | 1.69 [1 to 4]
  EORTCQLQ-C30 Post-transplant 11. Have you had trouble sleeping?: number analyzed (Participants) | 10 | 10
  EORTCQLQ-C30 Post-transplant 11. Have you had trouble sleeping? | 2.0 [1 to 4] | 1.6 [1 to 4]
  EORTCQLQ-C30 Screening 12. Have you felt weak?: number analyzed (Participants) | 22 | 25
  EORTCQLQ-C30 Screening 12. Have you felt weak? | 2.42 [1 to 4] | 2.04 [1 to 4]
  EORTCQLQ-C30 Pre-transplant 12. Have you felt weak?: number analyzed (Participants) | 14 | 13
  EORTCQLQ-C30 Pre-transplant 12. Have you felt weak? | 1.85 [1 to 4] | 1.77 [1 to 4]
  EORTCQLQ-C30 Post-transplant 12. Have you felt weak?: number analyzed (Participants) | 10 | 10
  EORTCQLQ-C30 Post-transplant 12. Have you felt weak? | 2.1 [1 to 4] | 1.7 [1 to 4]
  EORTCQLQ-C30 Screening 13. Have you lacked appetite?: number analyzed (Participants) | 22 | 25
  EORTCQLQ-C30 Screening 13. Have you lacked appetite? | 1.54 [1 to 4] | 1.72 [1 to 4]
  EORTCQLQ-C30 Pre-transplant 13. Have you lacked appetite?: number analyzed (Participants) | 14 | 13
  EORTCQLQ-C30 Pre-transplant 13. Have you lacked appetite? | 1.71 [1 to 4] | 1.85 [1 to 4]
  EORTCQLQ-C30 Post-transplant 13. Have you lacked appetite?: number analyzed (Participants) | 10 | 10
  EORTCQLQ-C30 Post-transplant 13. Have you lacked appetite? | 1.5 [1 to 4] | 1.70 [1 to 4]
  EORTCQLQ-C30 Screening 14. Have you felt nauseated?: number analyzed (Participants) | 22 | 25
  EORTCQLQ-C30 Screening 14. Have you felt nauseated? | 1.31 [1 to 4] | 1.4 [1 to 4]
  EORTCQLQ-C30 Pre-transplant 14. Have you felt nauseated?: number analyzed (Participants) | 14 | 13
  EORTCQLQ-C30 Pre-transplant 14. Have you felt nauseated? | 1.07 [1 to 4] | 1.53 [1 to 4]
  EORTCQLQ-C30 Post-transplant 14. Have you felt nauseated?: number analyzed (Participants) | 10 | 10
  EORTCQLQ-C30 Post-transplant 14. Have you felt nauseated? | 1.5 [1 to 4] | 1.4 [1 to 4]
  EORTCQLQ-C30 Screening 15. Have you vomited?: number analyzed (Participants) | 22 | 25
  EORTCQLQ-C30 Screening 15. Have you vomited? | 1.09 [1 to 4] | 1.12 [1 to 4]
  EORTCQLQ-C30 Pre-transplant 15. Have you vomited?: number analyzed (Participants) | 14 | 13
  EORTCQLQ-C30 Pre-transplant 15. Have you vomited? | 1 [1 to 4] | 1.08 [1 to 4]
  EORTCQLQ-C30 Post-transplant 15. Have you vomited?: number analyzed (Participants) | 10 | 10
  EORTCQLQ-C30 Post-transplant 15. Have you vomited? | 1.1 [1 to 4] | 1.1 [1 to 4]
  EORTCQLQ-C30 Screening 16. Have you been constipated?: number analyzed (Participants) | 22 | 25
  EORTCQLQ-C30 Screening 16. Have you been constipated? | 1.31 [1 to 4] | 1.52 [1 to 4]
  EORTCQLQ-C30 Pre-transplant 16. Have you been constipated?: number analyzed (Participants) | 14 | 13
  EORTCQLQ-C30 Pre-transplant 16. Have you been constipated? | 1.21 [1 to 4] | 1.38 [1 to 4]
  EORTCQLQ-C30 Post-transplant 16. Have you been constipated?: number analyzed (Participants) | 10 | 10
  EORTCQLQ-C30 Post-transplant 16. Have you been constipated? | 1 [1 to 4] | 1 [1 to 4]
  EORTCQLQ-C30 Screening 17. Have you had diarrhea?: number analyzed (Participants) | 22 | 25
  EORTCQLQ-C30 Screening 17. Have you had diarrhea? | 1.45 [1 to 4] | 1.20 [1 to 4]
  EORTCQLQ-C30 Pre-transplant 17. Have you had diarrhea?: number analyzed (Participants) | 14 | 13
  EORTCQLQ-C30 Pre-transplant 17. Have you had diarrhea? | 1.23 [1 to 4] | 1.23 [1 to 4]
  EORTCQLQ-C30 Post-transplant 17. Have you had diarrhea?: number analyzed (Participants) | 10 | 10
  EORTCQLQ-C30 Post-transplant 17. Have you had diarrhea? | 2.0 [1 to 4] | 1.5 [1 to 4]
  EORTCQLQ-C30 Screening 18. Were you tired?: number analyzed (Participants) | 22 | 25
  EORTCQLQ-C30 Screening 18. Were you tired? | 2.45 [1 to 4] | 2.4 [1 to 4]
  EORTCQLQ-C30 Pre-transplant 18. Were you tired?: number analyzed (Participants) | 14 | 13
  EORTCQLQ-C30 Pre-transplant 18. Were you tired? | 2.23 [1 to 4] | 2.31 [1 to 4]
  EORTCQLQ-C30 Post-transplant 18. Were you tired? | 2.10 [1 to 4] | 2.20 [1 to 4]
  EORTCQLQ-C30 Screening 19. Did pain interfere with your daily activities?: number analyzed (Participants) | 22 | 25
  EORTCQLQ-C30 Screening 19. Did pain interfere with your daily activities? | 1.27 [1 to 4] | 1.48 [1 to 4]
  EORTCQLQ-C30 Pre-transplant 19. Did pain interfere with your daily activities?: number analyzed (Participants) | 14 | 13
  EORTCQLQ-C30 Pre-transplant 19. Did pain interfere with your daily activities? | 1.61 [1 to 4] | 1.38 [1 to 4]
  EORTCQLQ-C30 Post-transplant 19. Did pain interfere with your daily activities?: number analyzed (Participants) | 10 | 10
  EORTCQLQ-C30 Post-transplant 19. Did pain interfere with your daily activities? | 1.5 [1 to 4] | 1.4 [1 to 4]
  EORTCQLQ-C30 Screening 20. Difficulty concentrating on things like reading a or watching TV?: number analyzed (Participants) | 22 | 25
  EORTCQLQ-C30 Screening 20. Difficulty concentrating on things like reading a or watching TV? | 1.81 [1 to 4] | 1.32 [1 to 4]
  EORTCQLQ-C30 Pre-transplant 20. Difficulty concentrating on things like reading a or watching TV?: number analyzed (Participants) | 14 | 13
  EORTCQLQ-C30 Pre-transplant 20. Difficulty concentrating on things like reading a or watching TV? | 1.69 [1 to 4] | 1.30 [1 to 4]
  EORTCQLQ-C30 Post-transplant 20. Difficulty concentrating on things like reading a or watching TV?: number analyzed (Participants) | 10 | 25
  EORTCQLQ-C30 Post-transplant 20. Difficulty concentrating on things like reading a or watching TV? | 1.3 [1 to 4] | 1.2 [1 to 4]
  EORTCQLQ-C30 Screening 21. Did you feel tense?: number analyzed (Participants) | 22 | 25
  EORTCQLQ-C30 Screening 21. Did you feel tense? | 1.72 [1 to 4] | 1.60 [1 to 4]
  EORTCQLQ-C30 pre-transplant 21. Did you feel tense?: number analyzed (Participants) | 14 | 13
  EORTCQLQ-C30 pre-transplant 21. Did you feel tense? | 1.92 [1 to 4] | 1.31 [1 to 4]
  EORTCQLQ-C30 Post-transplant 21. Did you feel tense?: number analyzed (Participants) | 10 | 10
  EORTCQLQ-C30 Post-transplant 21. Did you feel tense? | 1.5 [1 to 4] | 1.4 [1 to 4]
  EORTCQLQ-C30 Screening 22. Did you worry?: number analyzed (Participants) | 22 | 25
  EORTCQLQ-C30 Screening 22. Did you worry? | 2.13 [1 to 4] | 1.68 [1 to 4]
  EORTCQLQ-C30 Pre-transplant 22. Did you worry?: number analyzed (Participants) | 14 | 13
  EORTCQLQ-C30 Pre-transplant 22. Did you worry? | 2.0 [1 to 4] | 1.92 [1 to 4]
  EORTCQLQ-C30 Post-transplant 22. Did you worry?: number analyzed (Participants) | 10 | 10
  EORTCQLQ-C30 Post-transplant 22. Did you worry? | 1.8 [1 to 4] | 1.7 [1 to 4]
  EORTCQLQ-C30 Screening 23. Did you feel irritable?: number analyzed (Participants) | 22 | 25
  EORTCQLQ-C30 Screening 23. Did you feel irritable? | 1.63 [1 to 4] | 1.41 [1 to 4]
  EORTCQLQ-C30 Pre-Transplant 23. Did you feel irritable?: number analyzed (Participants) | 14 | 13
  EORTCQLQ-C30 Pre-Transplant 23. Did you feel irritable? | 1.77 [1 to 4] | 1.54 [1 to 4]
  EORTCQLQ-C30 Post-Transplant 23. Did you feel irritable?: number analyzed (Participants) | 10 | 10
  EORTCQLQ-C30 Post-Transplant 23. Did you feel irritable? | 1.7 [1 to 4] | 1.6 [1 to 4]
  EORTCQLQ-C30 Screening 24. Did you feel depressed?: number analyzed (Participants) | 22 | 25
  EORTCQLQ-C30 Screening 24. Did you feel depressed? | 1.68 [1 to 4] | 1.48 [1 to 4]
  EORTCQLQ-C30 Pre-Transplant 24. Did you feel depressed?: number analyzed (Participants) | 14 | 13
  EORTCQLQ-C30 Pre-Transplant 24. Did you feel depressed? | 1.41 [1 to 4] | 1.46 [1 to 4]
  EORTCQLQ-C30 Post-Transplant 24. Did you feel depressed?: number analyzed (Participants) | 10 | 10
  EORTCQLQ-C30 Post-Transplant 24. Did you feel depressed? | 1.5 [1 to 4] | 1.5 [1 to 4]
  EORTCQLQ-C30 Screening 25. Have you had difficulty remembering things?: number analyzed (Participants) | 22 | 25
  EORTCQLQ-C30 Screening 25. Have you had difficulty remembering things? | 1.86 [1 to 4] | 1.60 [1 to 4]
  EORTCQLQ-C30 Pre-transplant 25. Have you had difficulty remembering things?: number analyzed (Participants) | 14 | 13
  EORTCQLQ-C30 Pre-transplant 25. Have you had difficulty remembering things? | 1.84 [1 to 4] | 1.54 [1 to 4]
  EORTCQLQ-C30 Post-transplant 25. Have you had difficulty remembering things?: number analyzed (Participants) | 10 | 10
  EORTCQLQ-C30 Post-transplant 25. Have you had difficulty remembering things? | 1.9 [1 to 4] | 1.6 [1 to 4]
  EORTCQLQ-C30 Screening 26. Has your physical condition/medical treatment interfere with family?: number analyzed (Participants) | 22 | 25
  EORTCQLQ-C30 Screening 26. Has your physical condition/medical treatment interfere with family? | 1.90 [1 to 4] | 1.48 [1 to 4]
  EORTCQLQ-C30 Pre-transplant 26.Has your physical condition/medical treatment interfere w/family?: number analyzed (Participants) | 14 | 13
  EORTCQLQ-C30 Pre-transplant 26.Has your physical condition/medical treatment interfere w/family? | 2.15 [1 to 4] | 2.07 [1 to 4]
  EORTCQLQ-C30 Post-transplant 26.Has your physical condition/medical treatment interfere w/family?: number analyzed (Participants) | 10 | 10
  EORTCQLQ-C30 Post-transplant 26.Has your physical condition/medical treatment interfere w/family? | 1.8 [1 to 4] | 1.7 [1 to 4]
  EORTCQLQ-C30 Screening 27.Has your physical condition/medical treatment interfere w/social life?: number analyzed (Participants) | 22 | 25
  EORTCQLQ-C30 Screening 27.Has your physical condition/medical treatment interfere w/social life? | 2.09 [1 to 4] | 1.92 [1 to 4]
  EORTCQLQ-C30Pre-transplant 27.Has your physical condition/medical treatment interfere w/social life?: number analyzed (Participants) | 14 | 13
  EORTCQLQ-C30Pre-transplant 27.Has your physical condition/medical treatment interfere w/social life? | 2.5 [1 to 4] | 2.38 [1 to 4]
  EORTCQLQ-C30 Post-trans 27.Has your physical condition/medical treatment interfere w/social life?: number analyzed (Participants) | 10 | 10
  EORTCQLQ-C30 Post-trans 27.Has your physical condition/medical treatment interfere w/social life? | 2.1 [1 to 4] | 2.5 [1 to 4]
  EORTCQLQ-C30 Screening 28.Physical condition/medical treatment caused financial difficulties?: number analyzed (Participants) | 22 | 25
  EORTCQLQ-C30 Screening 28.Physical condition/medical treatment caused financial difficulties? | 1.71 [1 to 4] | 1.56 [1 to 4]
  EORTCQLQ-C30 Pre-transplant 28.Physical condition/medical treatment caused financial difficulties?: number analyzed (Participants) | 14 | 13
  EORTCQLQ-C30 Pre-transplant 28.Physical condition/medical treatment caused financial difficulties? | 2.38 [1 to 4] | 1.92 [1 to 4]
  EORTCQLQ-C30 Posttransplant 28.Physical condition/medical treatment caused financial difficulties?: number analyzed (Participants) | 10 | 10
  EORTCQLQ-C30 Posttransplant 28.Physical condition/medical treatment caused financial difficulties? | 2.0 [1 to 4] | 2.0 [1 to 4]
  EORTCQLQ-C30 Screening 29.How would you rate your overall health during the past week?: number analyzed (Participants) | 22 | 25
  EORTCQLQ-C30 Screening 29.How would you rate your overall health during the past week? | 4.52 [1 to 7] | 4.86 [1 to 7]
  EORTCQLQ-C30 Pre-transplant 29.How would you rate your overall health during the past week?: number analyzed (Participants) | 14 | 13
  EORTCQLQ-C30 Pre-transplant 29.How would you rate your overall health during the past week? | 4.77 [1 to 7] | 4.61 [1 to 7]
  EORTCQLQ-C30 Post-transplant 29.How would you rate your overall health during the past week?: number analyzed (Participants) | 10 | 10
  EORTCQLQ-C30 Post-transplant 29.How would you rate your overall health during the past week? | 5.4 [1 to 7] | 5.1 [1 to 7]
  EORTCQLQ-C30 Screening 30. How would you rate your overall quality of life during the past week?: number analyzed (Participants) | 22 | 25
  EORTCQLQ-C30 Screening 30. How would you rate your overall quality of life during the past week? | 4.5 [1 to 7] | 5.12 [1 to 7]
  EORTCQLQ-C30 Pretransplant 30.How would you rate your overall quality of life during the past week?: number analyzed (Participants) | 14 | 13
  EORTCQLQ-C30 Pretransplant 30.How would you rate your overall quality of life during the past week? | 4.46 [1 to 7] | 4.69 [1 to 7]
  EORTCQLQ-C30 Posttransplant 30.How would you rate your overall QoL during the past week?: number analyzed (Participants) | 10 | 10
  EORTCQLQ-C30 Posttransplant 30.How would you rate your overall QoL during the past week? | 5.1 [1 to 7] | 5.1 [1 to 7]

3. Secondary Outcome: Quality of Life Will be Assessed Using the EORTC QLQ-HDC29 a Supplementary Module Assessing the Quality of Life During and After High-dose Chemotherapy and Stem Cell Transplantation.
Description: European Organization for Research and Treatment of Cancer Quality of Life Questionnaire High Dose Chemotherapy (EORTC QLQ-HDC29) is a treatment-specific quality of life questionnaire that addresses treatment specific side effects as well as emotional, social, and family issues for patients treated with high dose regimens and HCT. The QLQ-HDC29 module includes 29 items, consisting of 6 multi-item scales and 8 single-items; all items employ a 4-point Likert scale, ranging from 1 (not at all) to 4 (very much) with lower scores representing a better outcome and higher scores a worse outcome with the exception of question 47 and 52 being the a higher score resulting in a better outcome and lower score a worse outcome.
Time Frame: EORTC QLQ-HDC29 questionnaire will be collected after completion of therapy (HMA 4-6 month, and up to 6 months for induction-like chemotherapy) pre stem cell infusion (HSCT), and 100 (± 14) days post stem cell infusion (HSCT).
Population: The QLQ-HDC29 is a validated and widely used questionnaire to assess QOL in cancer patients. For Arm A (Azacitidine or Decitabine) only 14 subjects submitted EORTC QLQ-HDC29 at pre-HCST and 10 subjects post-HSCT. For Arm B (induction chemo) 13 subjects submitted QLQ-HDC29 at pre-HSCT and 10 subjects post-HSCT. Scores for each question and timepoints were averaged to obtain mean. However, there are some questions were subjects noted N/A and these answered were subtracted from the number analyzed.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Arm A (Decitabine or Azacitidine) | Arm B (Induction-like Chemotherapy Regimen)
Number analyzed (Participants) | 25 | 25
units on a scale
  QLQ-HDC 29 Pre-HSCT 31. Have you had soreness in your mouth?: number analyzed (Participants) | 14 | 13
  QLQ-HDC 29 Pre-HSCT 31. Have you had soreness in your mouth? | 1.36 [1 to 4] | 1.08 [1 to 4]
  QLQ-HDC 29 Post-HSCT 31. Have you had soreness in your mouth?: number analyzed (Participants) | 10 | 10
  QLQ-HDC 29 Post-HSCT 31. Have you had soreness in your mouth? | 1.2 [1 to 4] | 1.0 [1 to 4]
  QLQ-HDC 29 Pre-HSCT 32. Have you had a dry mouth?: number analyzed (Participants) | 14 | 13
  QLQ-HDC 29 Pre-HSCT 32. Have you had a dry mouth? | 1.36 [1 to 4] | 1.62 [1 to 4]
  QLQ-HDC 29 Post-HSCT 32. Have you had a dry mouth?: number analyzed (Participants) | 10 | 10
  QLQ-HDC 29 Post-HSCT 32. Have you had a dry mouth? | 2.0 [1 to 4] | 1.7 [1 to 4]
  QLQ-HDC 29 Pre-HSCT 33. Have you had trouble swallowing?: number analyzed (Participants) | 14 | 13
  QLQ-HDC 29 Pre-HSCT 33. Have you had trouble swallowing? | 1.07 [1 to 4] | 1.15 [1 to 4]
  QLQ-HDC 29 Post-HSCT 33. Have you had trouble swallowing?: number analyzed (Participants) | 10 | 10
  QLQ-HDC 29 Post-HSCT 33. Have you had trouble swallowing? | 1.2 [1 to 4] | 1.3 [1 to 4]
  QLQ-HDC 29 Pre-HSCT 34. Did food and drink taste different from usual?: number analyzed (Participants) | 14 | 13
  QLQ-HDC 29 Pre-HSCT 34. Did food and drink taste different from usual? | 1.57 [1 to 4] | 1.92 [1 to 4]
  QLQ-HDC 29 Post-HSCT 34. Did food and drink taste different from usual?: number analyzed (Participants) | 10 | 10
  QLQ-HDC 29 Post-HSCT 34. Did food and drink taste different from usual? | 1.9 [1 to 4] | 2.2 [1 to 4]
  QLQ-HDC 29 Pre-HSCT 35. Have you had abdominal pains or cramps?: number analyzed (Participants) | 14 | 13
  QLQ-HDC 29 Pre-HSCT 35. Have you had abdominal pains or cramps? | 1.21 [1 to 4] | 1.38 [1 to 4]
  QLQ-HDC 29 Post-HSCT 35. Have you had abdominal pains or cramps?: number analyzed (Participants) | 10 | 10
  QLQ-HDC 29 Post-HSCT 35. Have you had abdominal pains or cramps? | 1.3 [1 to 4] | 1.6 [1 to 4]
  QLQ-HDC 29 Pre-HSCT 36. Have you had skin problems?: number analyzed (Participants) | 14 | 13
  QLQ-HDC 29 Pre-HSCT 36. Have you had skin problems? | 1.71 [1 to 4] | 1.38 [1 to 4]
  QLQ-HDC 29 Post-HSCT 36. Have you had skin problems?: number analyzed (Participants) | 10 | 10
  QLQ-HDC 29 Post-HSCT 36. Have you had skin problems? | 1.6 [1 to 4] | 1.5 [1 to 4]
  QLQ-HDC 29 Pre-HSCT 37. Have you been upset by how the treatment has affected your hair?: number analyzed (Participants) | 14 | 13
  QLQ-HDC 29 Pre-HSCT 37. Have you been upset by how the treatment has affected your hair? | 1.43 [1 to 4] | 1.38 [1 to 4]
  QLQ-HDC 29 Post-HSCT 37. Have you been upset by how the treatment has affected your hair?: number analyzed (Participants) | 10 | 10
  QLQ-HDC 29 Post-HSCT 37. Have you been upset by how the treatment has affected your hair? | 2.0 [1 to 4] | 1.7 [1 to 4]
  QLQ-HDC 29 Pre-HSCT 38. Have you worried about your weight being too low?: number analyzed (Participants) | 14 | 13
  QLQ-HDC 29 Pre-HSCT 38. Have you worried about your weight being too low? | 1.5 [1 to 4] | 1.62 [1 to 4]
  QLQ-HDC 29 Post-HSCT 38. Have you worried about your weight being too low?: number analyzed (Participants) | 10 | 10
  QLQ-HDC 29 Post-HSCT 38. Have you worried about your weight being too low? | 1.6 [1 to 4] | 2.2 [1 to 4]
  QLQ-HDC 29 Pre-HSCT 39. Have you had fevers or chills?: number analyzed (Participants) | 14 | 13
  QLQ-HDC 29 Pre-HSCT 39. Have you had fevers or chills? | 1.43 [1 to 4] | 1.46 [1 to 4]
  QLQ-HDC 29 Post-HSCT 39. Have you had fevers or chills?: number analyzed (Participants) | 10 | 10
  QLQ-HDC 29 Post-HSCT 39. Have you had fevers or chills? | 1.3 [1 to 4] | 1 [1 to 4]
  QLQ-HDC 29 Pre-HSCT 40. Did you urinate frequently?: number analyzed (Participants) | 14 | 13
  QLQ-HDC 29 Pre-HSCT 40. Did you urinate frequently? | 2.29 [1 to 4] | 2.0 [1 to 4]
  QLQ-HDC 29 Post-HSCT 40. Did you urinate frequently?: number analyzed (Participants) | 10 | 10
  QLQ-HDC 29 Post-HSCT 40. Did you urinate frequently? | 2.1 [1 to 4] | 1.4 [1 to 4]
  QLQ-HDC 29 Pre-HSCT 41. Have you had aches or pains in your bones?: number analyzed (Participants) | 14 | 13
  QLQ-HDC 29 Pre-HSCT 41. Have you had aches or pains in your bones? | 1.79 [1 to 4] | 1.46 [1 to 4]
  QLQ-HDC 29 Post-HSCT 41. Have you had aches or pains in your bones?: number analyzed (Participants) | 10 | 10
  QLQ-HDC 29 Post-HSCT 41. Have you had aches or pains in your bones? | 1.7 [1 to 4] | 1.4 [1 to 4]
  QLQ-HDC 29 Pre-HSCT 42. Have you found it difficult to finish things you started? | 1.64 [1 to 4] | 1.46 [1 to 4]
  QLQ-HDC 29 Post-HSCT 42. Have you found it difficult to finish things you started?: number analyzed (Participants) | 10 | 10
  QLQ-HDC 29 Post-HSCT 42. Have you found it difficult to finish things you started? | 1.6 [1 to 4] | 1.3 [1 to 4]
  QLQ-HDC 29 Pre-HSCT 43. Did you worry about the results of examinations and tests?: number analyzed (Participants) | 14 | 13
  QLQ-HDC 29 Pre-HSCT 43. Did you worry about the results of examinations and tests? | 1.92 [1 to 4] | 1.66 [1 to 4]
  QLQ-HDC 29 Post-HSCT 43. Did you worry about the results of examinations and tests?: number analyzed (Participants) | 10 | 10
  QLQ-HDC 29 Post-HSCT 43. Did you worry about the results of examinations and tests? | 1.7 [1 to 4] | 1.7 [1 to 4]
  QLQ-HDC 29 Pre-HSCT 44. Have you had trouble coping with the hospital stay?: number analyzed (Participants) | 5 | 6
  QLQ-HDC 29 Pre-HSCT 44. Have you had trouble coping with the hospital stay? | 1.6 [1 to 4] | 1.5 [1 to 4]
  QLQ-HDC 29 Post-HSCT 44. Have you had trouble coping with the hospital stay?: number analyzed (Participants) | 2 | 3
  QLQ-HDC 29 Post-HSCT 44. Have you had trouble coping with the hospital stay? | 1.0 [1 to 4] | 1.0 [1 to 4]
  QLQ-HDC 29 Pre-HSCT 45. Has the isolation in the hospital troubled you?: number analyzed (Participants) | 3 | 6
  QLQ-HDC 29 Pre-HSCT 45. Has the isolation in the hospital troubled you? | 1.66 [1 to 4] | 1.66 [1 to 4]
  QLQ-HDC 29 Post-HSCT 45. Has the isolation in the hospital troubled you?: number analyzed (Participants) | 2 | 3
  QLQ-HDC 29 Post-HSCT 45. Has the isolation in the hospital troubled you? | 1.0 [1 to 4] | 1.0 [1 to 4]
  QLQ-HDC 29 Pre-HSCT 46. Have you worried that the blood counts may not recover?: number analyzed (Participants) | 3 | 6
  QLQ-HDC 29 Pre-HSCT 46. Have you worried that the blood counts may not recover? | 2.0 [1 to 4] | 1.83 [1 to 4]
  QLQ-HDC 29 Post-HSCT 46. Have you worried that the blood counts may not recover?: number analyzed (Participants) | 2 | 3
  QLQ-HDC 29 Post-HSCT 46. Have you worried that the blood counts may not recover? | 1.5 [1 to 4] | 3.33 [1 to 4]
  QLQ-HDC 29 Pre-HSCT 47. How satisfied were you with the preparation for your treatment?: number analyzed (Participants) | 3 | 6
  QLQ-HDC 29 Pre-HSCT 47. How satisfied were you with the preparation for your treatment? | 2.33 [1 to 4] | 2.83 [1 to 4]
  QLQ-HDC 29 Post-HSCT 47. How satisfied were you with the preparation for your treatment?: number analyzed (Participants) | 2 | 2
  QLQ-HDC 29 Post-HSCT 47. How satisfied were you with the preparation for your treatment? | 2.5 [1 to 4] | 2.5 [1 to 4]
  QLQ-HDC 29 Pre-HSCT 48. Have you felt isolated from those close to you (family, friends)?: number analyzed (Participants) | 14 | 13
  QLQ-HDC 29 Pre-HSCT 48. Have you felt isolated from those close to you (family, friends)? | 1.77 [1 to 4] | 1.77 [1 to 4]
  QLQ-HDC 29 Post-HSCT 48. Have you felt isolated from those close to you (family, friends)?: number analyzed (Participants) | 10 | 10
  QLQ-HDC 29 Post-HSCT 48. Have you felt isolated from those close to you (family, friends)? | 1.7 [1 to 4] | 1.6 [1 to 4]
  QLQ-HDC 29 Pre-HSCT49.Have you been concerned about disruption to your family life due to treatment?: number analyzed (Participants) | 14 | 13
  QLQ-HDC 29 Pre-HSCT49.Have you been concerned about disruption to your family life due to treatment? | 1.92 [1 to 4] | 2.23 [1 to 4]
  QLQ-HDC29Post HSCT 49.Have you been concerned about disruption to your family life due to treatment?: number analyzed (Participants) | 10 | 10
  QLQ-HDC29Post HSCT 49.Have you been concerned about disruption to your family life due to treatment? | 1.5 [1 to 4] | 2.22 [1 to 4]
  QLQ-HDC29 Pre HSCT 50. How distressing do you think your illness/treatment has been to those close?: number analyzed (Participants) | 14 | 13
  QLQ-HDC29 Pre HSCT 50. How distressing do you think your illness/treatment has been to those close? | 2.62 [1 to 4] | 2.69 [1 to 4]
  QLQ-HDC29 Post-HSCT 50. How distressing do you think your illness/treatment has been to those close?: number analyzed (Participants) | 10 | 10
  QLQ-HDC29 Post-HSCT 50. How distressing do you think your illness/treatment has been to those close? | 2.6 [1 to 4] | 2.5 [1 to 4]
  QLQ-HDC29 Pre-HSCT 51. Have you felt a need to keep fears/concerns from family or friends?: number analyzed (Participants) | 14 | 13
  QLQ-HDC29 Pre-HSCT 51. Have you felt a need to keep fears/concerns from family or friends? | 1.62 [1 to 4] | 1.84 [1 to 4]
  QLQ-HDC29 Post-HSCT 51. Have you felt a need to keep fears/concerns from family or friends?: number analyzed (Participants) | 10 | 10
  QLQ-HDC29 Post-HSCT 51. Have you felt a need to keep fears/concerns from family or friends? | 1.8 [1 to 4] | 2.2 [1 to 4]
  Pre-HSCT 52.Has your experience helped u distinguish between important/non-important things in life?: number analyzed (Participants) | 12 | 13
  Pre-HSCT 52.Has your experience helped u distinguish between important/non-important things in life? | 2.83 [1 to 4] | 2.54 [1 to 4]
  PostHSCT 52.Has your experience helped u distinguish between important/non-important things in life?: number analyzed (Participants) | 10 | 10
  PostHSCT 52.Has your experience helped u distinguish between important/non-important things in life? | 2.1 [1 to 4] | 3.1 [1 to 4]
  QLQ-HDC29 Pre-HSCT 53. Were you worried about your health in the future?: number analyzed (Participants) | 13 | 13
  QLQ-HDC29 Pre-HSCT 53. Were you worried about your health in the future? | 2.23 [1 to 4] | 2.46 [1 to 4]
  QLQ-HDC29 Post-HSCT 53. Were you worried about your health in the future?: number analyzed (Participants) | 10 | 10
  QLQ-HDC29 Post-HSCT 53. Were you worried about your health in the future? | 2.5 [1 to 4] | 2.5 [1 to 4]
  QLQ-HDC29 Pre-HSCT 54. Have you felt physically less attractive due to illness/treatment?: number analyzed (Participants) | 13 | 13
  QLQ-HDC29 Pre-HSCT 54. Have you felt physically less attractive due to illness/treatment? | 2.0 [1 to 4] | 1.92 [1 to 4]
  QLQ-HDC29 Post-HSCT 54. Have you felt physically less attractive due to illness/treatment?: number analyzed (Participants) | 10 | 10
  QLQ-HDC29 Post-HSCT 54. Have you felt physically less attractive due to illness/treatment? | 2.4 [1 to 4] | 2.1 [1 to 4]
  QLQ-HDC29 Pre-HSCT 55. Have you been concerned about your ability to have children?: number analyzed (Participants) | 4 | 4
  QLQ-HDC29 Pre-HSCT 55. Have you been concerned about your ability to have children? | 1.75 [1 to 4] | 1.25 [1 to 4]
  QLQ-HDC29 Post-HSCT 55. Have you been concerned about your ability to have children?: number analyzed (Participants) | 3 | 1
  QLQ-HDC29 Post-HSCT 55. Have you been concerned about your ability to have children? | 1.33 [1 to 4] | 1 [1 to 4]
  QLQ-HDC29 Pre-HSCT 56. Did having to take your drugs regularly interfere with your daily life?: number analyzed (Participants) | 7 | 9
  QLQ-HDC29 Pre-HSCT 56. Did having to take your drugs regularly interfere with your daily life? | 1.28 [1 to 4] | 1.88 [1 to 4]
  QLQ-HDC29 Post-HSCT 56. Did having to take your drugs regularly interfere with your daily life?: number analyzed (Participants) | 10 | 9
  QLQ-HDC29 Post-HSCT 56. Did having to take your drugs regularly interfere with your daily life? | 1.9 [1 to 4] | 2.11 [1 to 4]
  QLQ-HDC29 Pre-HSCT 57. Have you been watching yourself closely for any new symptoms?: number analyzed (Participants) | 6 | 9
  QLQ-HDC29 Pre-HSCT 57. Have you been watching yourself closely for any new symptoms? | 2.66 [1 to 4] | 2.77 [1 to 4]
  QLQ-HDC29 Post-HSCT 57. Have you been watching yourself closely for any new symptoms?: number analyzed (Participants) | 10 | 9
  QLQ-HDC29 Post-HSCT 57. Have you been watching yourself closely for any new symptoms? | 3.3 [1 to 4] | 3.66 [1 to 4]
  QLQ-HDC29 Pre-HSCT 58. Have you felt less interest in sex?: number analyzed (Participants) | 6 | 9
  QLQ-HDC29 Pre-HSCT 58. Have you felt less interest in sex? | 2.33 [1 to 4] | 2.55 [1 to 4]
  QLQ-HDC29 Post-HSCT 58. Have you felt less interest in sex?: number analyzed (Participants) | 10 | 8
  QLQ-HDC29 Post-HSCT 58. Have you felt less interest in sex? | 2.50 [1 to 4] | 2.25 [1 to 4]
  QLQ-HDC29 Pre-HSCT 59. Have you felt less sexual enjoyment?: number analyzed (Participants) | 6 | 9
  QLQ-HDC29 Pre-HSCT 59. Have you felt less sexual enjoyment? | 2.16 [1 to 4] | 2.66 [1 to 4]
  QLQ-HDC29 Post-HSCT 59. Have you felt less sexual enjoyment?: number analyzed (Participants) | 10 | 8
  QLQ-HDC29 Post-HSCT 59. Have you felt less sexual enjoyment? | 2.6 [1 to 4] | 2.25 [1 to 4]

4. Secondary Outcome: Overall Survival
Description: The total length of follow-up will be 18 months from the start of treatment (day 1). Four categories were added for participants alive 18 months from start of treatment (day 1) 1) Participants alive after 18 months from start of treatment who received hematopoietic cell transplantation (HCT); 2) Participants alive after 18months from start of treatment who did not receive HCT.; 3) Participants deceased after 18 months from start of treatment who received HCT; 4) Participants deceased after 18 months from start of treatment who did not receive HCT.
Time Frame: Up to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Decitabine or Azacitidine) | Arm B (Induction-like Chemotherapy Regimen)
Number analyzed (Participants) | 25 | 25
Participants
  Participants alive after 18 months from start of treatment who received HCT. | 7 | 10
  Participants alive after 18months from start of treatment who did not receive HCT. | 2 | 1
  Participants deceased after 18 months from start of treatment who received HCT. | 5 | 3
  Participants deceased after 18 months from start of treatment who did not receive HCT. | 11 | 11

5. Secondary Outcome: Number of Patients Who Relapse Post-transplant
Description: To compare which of the two, intensive chemotherapy versus hypomethylating agent-based therapy, have a factor of relapse post hematopoietic cell transplantation (HCT).
Time Frame: Up to 18 months
Population: Only participants who received a HCT that relapse were assessed for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Decitabine or Azacitidine) | Arm B (Induction-like Chemotherapy Regimen)
Number analyzed (Participants) | 12 | 13
Participants
  Relapse post HCT | 6 | 3
  Did not relapse post HCT | 6 | 10

6. Secondary Outcome: Number of Participants Who Received a Hematopoietic Cell Transplantation (HCT).
Description: Frequency at which the participants received a hematopoietic cell transplantation (HCT)
Time Frame: Up to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Decitabine or Azacitidine) | Arm B (Induction-like Chemotherapy Regimen)
Number analyzed (Participants) | 25 | 25
Participants
  Received hematopoietic cell transplantation | 12 | 13
  Did not receive hematopoietic cell transplantation | 13 | 12

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was assessed up to 18 months from start of treatment.
Description: Serious AEs and Other AEs were not collected for this study. Only All-Cause Mortality was monitored.
Arm/Group | Arm A (Decitabine or Azacitidine) | Arm B (Induction-like Chemotherapy Regimen)
All-Cause Mortality (participants affected / at risk) | 16/25 | 14/25
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/52/NCT01812252/Prot_SAP_000.pdf